CLINICAL TRIAL: NCT01986335
Title: Phase 3 of Protectivity and Safety of DTP/HB/Hib (Bio Farma) Vaccines in Infants, Batch Consistency, Multi Center Trial
Brief Title: Protectivity and Safety of DTP/HB/Hib (Bio Farma) Vaccines in Infants, Batch Consistency, Multi Center Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Penta 0312
Record Dates: First submitted 2013-10-30; First posted 2013-11-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Combined pentavalent DTP/HB/Hib vaccine; Infants; Primary vaccination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DTP/HB/Hib Vaccine (Batch: A) (Experimental): Purified diphteria toxoid Purified tetanus toxoid Inactivated Bordetella pertussis HbsAg PRP-TT Aluminum phosphate Natrium Chloride Thimerosal
  Interventions: Biological: DTP/HB/Hib Vaccine
- DTP/HB/Hib vaccine (Batch: B) (Experimental): Purified diphteria toxoid Purified tetanus toxoid Inactivated Bordetella pertussis HbsAg PRP-TT Aluminum phosphate Natrium Chloride Thimerosal
  Interventions: Biological: DTP/HB/Hib Vaccine
- DTP/HB/Hib vaccine (Batch: C) (Experimental): Purified diphteria toxoid Purified tetanus toxoid Inactivated Bordetella pertussis HbsAg PRP-TT Aluminum phosphate Natrium Chloride Thimerosal
  Interventions: Biological: DTP/HB/Hib Vaccine

INTERVENTIONS:
Biological: DTP/HB/Hib Vaccine — DPT/HB/Hib vaccine (Bio Farma)
  Other Names: Pentavalent

SUMMARY:
The objectives of this study were to analyze the immunogenicity and reactogenicity of DTP/HB/Hib (Bio Farma) combination vaccine.

DETAILED DESCRIPTION:
This trial was randomized, double blind, prospective intervention and multi centers. Total 600 subject (6-11 weeks of ages) followed this trial, divided into 3 groups, each group consists of 200 subjects. A number of 342 subjects were recruited in Bandung, while 258 subjects were recruited in Jakarta.

ELIGIBILITY:
Inclusion Criteria:

* Infant 6-11 week of age
* Infant born after 37-42 week of pregnancy
* Infant weighting more than 2.5 kg at birth
* Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form
* Parents commit themselves to comply with the indication of the investigator and with the schedule of the trial
* Mother at least graduate from elementary school
* Received Hepatitis B vaccine (Bio Farma) at birth

Exclusion Criteria:

* Child concomitantly enroll or schedule to be enroll in another trial
* Evolving moderate or severe illness, especially infectious diseases or fever (axillary temperature >=37.5 Celsius on Day 0)
* Known history of allergy to any component of the vaccine component (e.g.formaldehyde)
* History of uncontrolled coagulopathy or blood disorder contraindicating intramuscular injection
* Known history of congenital or acquired immunodeficiency (including HIV infection)
* Child who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulin, blood derived product or long term corticotherapy (>2 weeks)
* Other vaccination within the 1 month prior to inclusion with the exception of BCG and poliomyelitis
* Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objective
* Infant with a known history of diphteria, tetanus, pertussis, Hib, Hepatitis B infection

Ages: 6 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Protectivity of DTP/HB/Hib (Bio Farma) vaccine | 4 months
  Number and percentage of infants with anti diphteria titer and anti tetanus titer >= 0.01 IU/ml, AntiHBs titer >=10mlIU/ml, and antiHib titer >= 0,15ug/ml 28 days after the last injection

SECONDARY OUTCOMES:
Antibody response to diphtheria between groups (three different batch numbers) | 4 months
  Serological response to Diphteria toxoid: GMT, percentage of infants with titer >=0.01 IU/ml and >=0.1 IU/ml, percentage of infants with increasing antibody titer >=4 times and/or percentage of infants with transition of seronegative to seropositive
Antibody response to Tetanus between groups (three different batch numbers) | 4 months
  Serological response to Tetanus toxoid: GMT, percentage of infants with titer >=0.01 IU/ml and >=0.1 IU/ml, percentage of infants with increasing antibody titer >=4 times and/or percentage of infants with transition of seronegative to seropositive
Antibody response to Pertussis component between groups (three different batch numbers) | 4 months
  Serological response to Pertussis component (agglutinins): GMT,percentage of infants with titre >=40, >=80,>=160 and >=320 (1/dil.), percentage of infants with increasing antibody titer >=4 times.
Antibody response to Hepatitis B between groups (three different batch numbers) | 4 months
  Serological response to Hepatitis B: Geometric mean of anti-HBs,percentage of infants with titer >=10mlIU/ml, percentage of infants with increasing antibody titer >=4 times and/ or percentage of infants with transition of seronegative to seropositive.
Antibody response to Hib/PRP between groups (three different batch numbers) | 4 months
  Serological response to Hib/PRP: GMT, percentage of infants with titre >=1ug/ml and >=0.15ug/ml, percentage of infants with increasing antibody titer >=4 times and/or percentage of infants with transition of seronegative to seropositive
Incidence rate of adverse event of DTP/HB/Hib (Bio Farma)vaccine between groups | 30 minutes, 72 hours, 28 days after immunization
  Number and percentage of local reaction and systemic events following vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Kusnandi Rusmil, PhD, Principal Investigator — Faculty of Medicine UNPAD; Hartono Gunardi, PhD, Principal Investigator — Faculty of Medicine UI
Locations (6):
- Indonesia (6):
  - Jatinegara Primary Health Center, Jakarta, Jakarta Special Capital Region
  - Mampang Prapatan Primary Health Center, Jakarta, Jakarta Special Capital Region
  - Tebet Primary Health Center, Jakarta, Jakarta Special Capital Region
  - Garuda Primary Health Center, Bandung, West Java
  - Ibrahim Adji Primary Health Center, Bandung, West Java
  - Puter Primary Health Center, Bandung, West Java

REFERENCES:
- [Derived] Rusmil K, Gunardi H, Fadlyana E, Soedjatmiko, Dhamayanti M, Sekartini R, Satari HI, Risan NA, Prasetio D, Tarigan R, Garheni R, Milanti M, Hadinegoro SR, Tanuwidjaja S, Bachtiar NS, Sari RM. The immunogenicity, safety, and consistency of an Indonesia combined DTP-HB-Hib vaccine in expanded program on immunization schedule. BMC Pediatr. 2015 Dec 19;15:219. doi: 10.1186/s12887-015-0525-2. PMID 26686508